CLINICAL TRIAL: NCT03638427
Title: Screening for Cervical Intraepithelial Neoplasia Using Self-collected Menstrual Blood
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul D Blumenthal, Professor, Stanford University
Other Study IDs: IRB-47250; NCI-2020-04139 (Registry Identifier: CTRP); GYNCVX0005 (Other: Stanford OnCore)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: HPV - Anogenital Human Papilloma Virus Infection
Keywords: menstrual blood, high risk HPV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High Risk HPV Positive Cohort: This group of women have tested positive for HR-HPV at annual cervical cancer screening and have been invited to participate in the study. They will be asked to use a menstrual pad we provide that collects a sample of their menstrual blood (strip). The strip will be mailed back to us for analysis (Menstrual Blood Analysis). These women will also be asked to conduct a self-swab vaginally to be sent back to us for analysis. These women will return 6-months after their positive HR-HPV for standard of care testing. All results of the standard of care tests, menstrual blood tests, and self-swab tests will be compared.
  Interventions: Diagnostic Test: Menstrual Blood Analysis (Menstrual Blood Analysis)

INTERVENTIONS:
Diagnostic Test: Menstrual Blood Analysis (Menstrual Blood Analysis) — We will be testing women's menstrual blood to investigate the feasibility and efficacy of assessing HR-HPV DNA and HPV E6/E7 mRNA via self-collected menstrual blood from a menstrual pad.

SUMMARY:
The purpose of this study is to investigate the feasibility and efficacy of assessing HR-HPV DNA and HPV E6/E7 mRNA via self-collected menstrual blood in a smart menstrual pad. In other words, can the investigators detect the high risk strains of the human papilloma virus (HPV) that are associated with cervical cancer in self-collected menstrual blood, as an alternative to collecting vaginal swabs.

ELIGIBILITY:
Inclusion Criteria:

There will be two study groups: 1) menstruating women over the age of 18 who have previous history of HR-HPV in the last 18 months and 2) menstruating women over the age of 18 who do not have a previous history of HR-HPV.

Exclusion Criteria:

* Women younger than 18 years old or are not menstruating regularly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Menstruating women over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Blumenthal, MD, MPH, Principal Investigator — Stanford University, Department of OB/GYN
Locations (1):
- Stanford Gynecology Clinic, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Naseri S, Young S, Cruz G, Blumenthal PD. Screening for High-Risk Human Papillomavirus Using Passive, Self-Collected Menstrual Blood. Obstet Gynecol. 2022 Sep 1;140(3):470-476. doi: 10.1097/AOG.0000000000004904. Epub 2022 Aug 3. PMID 35926207

RESULTS

PARTICIPANT FLOW:
Groups:
- High Risk HPV Positive Cohort: Testing of women's menstrual blood to investigate the feasibility and efficacy of assessing HR-HPV DNA and HPV E6/E7 mRNA self-collected via menstrual pad.
Period: Overall Study
Arm/Group | High Risk HPV Positive Cohort
Started | 159
Completed | 110
Not Completed | 49

BASELINE CHARACTERISTICS:
Arm/Group | High Risk HPV Positive Cohort
Number analyzed (Participants) | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 159
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 133
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 55
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 4
  White | 74
  More than one race | 3
  Unknown or Not Reported | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 159

OUTCOME MEASURES:

1. Primary Outcome: Agreement Between Modified Menstrual Pad and Clinician-Collected Specimen
Description: The clinician collected a vaginal swab to detect HPV, then participants used a modified menstrual pad to self-collect a sample within 2 months of the clinician collected swab (may have happened at up to 4 mo.). Participants may have had prior history of dysplasia or HPV positivity, or were from general population receiving regular check-up.
  Agreement between the clinician-collected swabs and participant-collected menstrual samples was assessed in:
  * Participants who sent their sample to the lab within 2 months, and whose sample was analyzed for the presence of HPV
  * Participants enrolled at the time of a previously scheduled colposcopy, with a biopsy taken (if clinically appropriate) showing moderate-to-severe dysplasia (cervical intraepithelial neoplasia [CIN] 2 or worse)
  * Participants enrolled at the time of a previously scheduled colposcopy, with a biopsy taken showing moderate-to-severe dysplasia, and participants whose laboratory results indicated presence of high-risk HPV.
Time Frame: 2-4-months after initial clinician collected samples were obtained and sent for HR-HPV DNA or HPV E6/E7 mRNA
Population: Participants with specimens meeting clinical criteria for each analysis category
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | High Risk HPV Positive Cohort
Number analyzed (Participants) | 46
percentage of agreement
  Participants who returned sample within 2 months | 93.5 [82.5 to 97.8]
  Participants with dysplasia CIN2 or worse: number analyzed (Participants) | 5
  Participants with dysplasia CIN2 or worse | 100 [32.5 to 100]
  Participants with dysplasia CIN2 worse and participants with lab results showing high-risk HPV: number analyzed (Participants) | 7
  Participants with dysplasia CIN2 worse and participants with lab results showing high-risk HPV | 100 [40.2 to 100]

2. Primary Outcome: Agreement Between Self-collected Vaginal Swabs vs Clinician-collected Cervical Specimens With High-risk HPV-Positive Results
Time Frame: 2-4-months after initial positive screen for HR-HPV DNA or HPV E6/E7 mRNA
Population: Participants with with high-risk HPV-positive results and who had cervical specimens collected
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | High Risk HPV Positive Cohort
Number analyzed (Participants) | 37
percentage of agreement | 88.1 [75.0 to 94.8]

3. Secondary Outcome: Number of Participants Who Preferred the Modified Menstrual Pad to Clinician-collected Cervical Specimens
Time Frame: 2-4-months after initial positive screen for HR-HPV DNA or HPV E6/E7 mRNA
Population: Participants who returned modified menstrual pads and indicated preference on exit survey
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk HPV Positive Cohort
Number analyzed (Participants) | 83
Participants | 78

4. Secondary Outcome: Number of Participants Who Opted Out of Self-swab Due to Discomfort With the Procedure
Time Frame: 2-4-months after initial positive screen for HR-HPV DNA or HPV E6/E7 mRNA
Population: Participants with available data
Measure: Count of Participants; unit: Participants
Arm/Group | High Risk HPV Positive Cohort
Number analyzed (Participants) | 141
Participants | 32

ADVERSE EVENTS:
Time Frame: On average up to 120 days
Arm/Group | High Risk HPV Positive Cohort
All-Cause Mortality (participants affected / at risk) | 0/159
Serious Adverse Events (participants affected / at risk) | 0/159
Other Adverse Events (participants affected / at risk) | 0/159

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT03638427/Prot_SAP_000.pdf